CLINICAL TRIAL: NCT06673550
Title: Fluid-filled Intragastric Balloon's Filling Volume At 500, 600, or 700 Ml for Treatment of Overweight and Obesity: Which is the Magic Number? a Single Centre Randomized Study
Brief Title: Intragastric Balloon for Treatment of Overweight and Obesity: Which is the Best Filling Volume?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mater Olbia Hospital (Other)
Responsible Party: Principal Investigator, Salvatore F. Vadalà di Prampero, MD, PhD, Mater Olbia Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001501/28/08/2024
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Obese Patients
Keywords: Intragastric balloon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fluid filled intragastric balloon at a volume of 500 ml (Experimental): This arm will undergo a fluid-filled intragastric balloon palcement at a volume of 500 ml
  Interventions: Procedure: Intragastric balloon
- Fluid filled intragastric balloon at a volume of 600 ml (Experimental): This arm will undergo a fluid-filled intragastric balloon palcement at a volume of 600 ml
  Interventions: Procedure: Intragastric balloon
- Fluid filled intragastric balloon at a volume of 700 ml (Experimental): This arm will undergo a fluid-filled intragastric balloon palcement at a volume of 700 ml
  Interventions: Procedure: Intragastric balloon

INTERVENTIONS:
Procedure: Intragastric balloon — Randomized trial comparing fluide-filled intragastric balloon at different filling volumes.

SUMMARY:
TITLE: Randomized study conducted in a single center, with the aim of comparing the three main filling volumes of the intragastric balloon in overweight or obese patients (BMI >27 and <60 kg/m2).

OBJECTIVE: To establish the efficacy and safety of the intragastric balloon inflated to different volumes in patients who are candidates for balloon placement for overweight or obesity. To date there is no well-defined filling volume and each Endoscopist inflates the balloon to a random volume between 500 and 700 ml according to the experience acquired, but without a clear rationale.

DESIGN: All overweight or obese patients with an indication for intragastric balloon placement will be preliminarily examined by a multidisciplinary team composed of a gastroeterologist, surgeon, nutritionist, psychologist, radiologist and endocrinologist.

Before each bariatric procedure, patients will undergo a psychometric and nutritional evaluation in order to identify any psychopathological conditions that contraindicate the operation.

The enrolled patients will be randomly divided to be candidates for balloon placement:

* 1/3 of patients will undergo treatment with an intragastric balloon inflated with 500 ml of saline solution and methylene blue, a space-occupying technique, which will be left in place for 1 year;
* 1/3 of patients will undergo treatment with an intragastric balloon inflated with 600 ml of saline solution and methylene blue;
* 1/3 of patients will undergo treatment with an intragastric balloon inflated with 700 ml of saline solution and methylene blue.

All balloons will remain in place for 6 months, as per the instructions provided in the product technical data sheet.

All the techniques described have already been widely validated by the scientific literature and are commonly used in bariatric endoscopy.

Sample size: assuming a significant level of 0.05, to detect as significant a medium effect size (f=0.25) with a power of 80% performing an ANOVA model we will need to enrol 156 patients (52 in each group). Taking into account a possible 5% of drop-out at the enrollment, the total number of patients will be around 165 (55 per group).

INFORMED CONSENT: Will be obtained upon first registration of the patient in the computer archive, as required by the hospital computer system, for access to personal data, which will be then used anonymously.

DETAILED DESCRIPTION:
INVESTIGATOR INITIATED STUDY A single-center, randomized study will be conducted in order to compare the three main fluid-filled intragastric balloon's (FF-IGB) filling volumes (500, 600 or 700 ml) for treatment of patients with overweight and obesity (BMI >27 and <60 kg/m2) at Gastroenterology and Gastrointestinal Endoscopy Unit, Mater Olbia Hospital, Qatar Foundation Endowment & Gemelli Foundation, Italy in period August 2022 - June 2025, with the aim to evaluate to assess efficacy and safety of different IGB volumes in our cohort.

BACKGROUND Obesity is now recognized as one of the most important public health issues. As excess weight continues to rise, its related comorbidities are also increasing and substantially impact on life expectancy. Population-based studies showed that trajectory of the obesity epidemic in the early childhood and adolescents is also increasing. The worldwide prevalence of excess weight in 1975 for girls was 0.7% and is calculated as 5.6% in 2016, and an increase from 0.9% to 7.8% in 2016 is reported for boys. Due to growing burden of obesity and associated complications there is an unmet need for therapeutical options than those currently available. As the sole nutritional and lifestyle modification is not sufficient in most cases, pharmacological or interventional procedural are often necessary. These led to rapid development of bariatric techniques that are evolving in the past decade . Endoscopic bariatric procedures are considered low-risk procedures and are applicable to the population who are not candidates for bariatric surgery. These procedures are combined with conservative measures for treatment of obesity and related co-morbidities. IGB placement is a bariatric procedure that involves insertion of a balloon in the stomach reducing its volume. They are usually filled with a fluid (saline solution, together with methylene blue) or, less frequently, with gas. IGB therapy effectively achieves short-term weight loss in obese patients in comparison to lifestyle modification alone. There is still no consensus on which is the best filling volume for IGB, that is usually filled according to the physician's expertise, with the aim to tailor the filling on patient's body mass index and stomach dimensions. This study aimed to evaluate weight loss and safety outcome after IGB and to analyze the difference between different filling volumes.

TYPE OF STUDY Single centre, randomized study.

OBJECTIVES The primary objective of the trial will be to compare three different filling volumes of IGB in the treatment of morbid obesity, with a hypothesis that percentage excess weight loss after IGB removal would be equivalent at a different filling volume. The secondary objective will be to test the possible differences between the different filling volumes regarding the percentage of adverse events (AEs), percentage of early IGB removal and quality of life (QOL).

ENDPOINTS Primary endpoint The primary end point will be weight loss defined by percentage of TWL (initial weight minus current weight) / (initial weight) x 100) and percentage EWL (initial weight minus follow-up weight) / (initial weight minus ideal weight for BMI 25) x 100%).

Secondary endpoints The secondary end points will include evaluation of adverse events (epigastric pain, nausea and vomiting, or any other issues (i.e., electrolyte imbalance, chest pain) requiring additional medical/endoscopic therapy or clinical investigation during hospitalization or until removal), detection of early removal, improvement of disease specific QOL measured by EQ-5D test

TRIAL DESIGN All patients with indication to FF-IGB will be revised by an internal multidisciplinary team composed of gastroenterologist, surgeon, dietitian, psychiatrist, radiologist and endocrinologist.

Before each endoscopic bariatric procedure, the patients will be subjected to a psychoclinical assessment (a clinical interview along with psychometric tests) to identify psychopathological conditions which may contraindicate the treatment or personality traits that may predict a successfull treatment (Millon Clinical Multiaxial Inventory-III, MCMI-III) ; during this visit it will be also evaluated the patients' food-related behavior (Eating Problem Checklist EPCL) , their binge eating severity (Binge Eating Scale BES) , various aspects of body-image perception and body attitudes (Body Uneasiness Test BUT), the eating impulsivity (BIS-11 Barratt Impulsiveness Scale BIS-11), and the patients' quality of life based on a combination of generic and specific instruments (Obesity Related Well-Being questionnaire ORWELL 97), collateral QoL measures (as the Short Form of SF-36 health Survey, SF-12 and BAROS Bariatric Analysis and Reporting Outcome System), together with the patients' own intervention; major endocrine disorders will be excluded.

Before each endoscopic bariatric procedure patients also will get an additional dietician examination while at hospital. During the first visit, all patients will be subjected to a clinical interview in order to estimate their calories intake, their eating and taste habits and their level of physical activity, then will be collected anthropometric data (height, weight, circumferences) in order to calculate Body Mass Index (BMI), Waist/Hips ratio (WHR) and cardiovascular risk. Furthermore, the dietician will identify a goal for each patient in terms of weight loss and physical activity improvement per week, reinforcing successful outcomes and rewarding good behaviors, also through the involvement of patients' family members as social support. Just after the endoscopic bariatric procedure patients will be given a two months refeeding protocol.

The patients undergoing the bariatric procedure will be randomly divided as follows:

* 1/3 patients will be treated with fluid-filled IGB inflated with 500 ml of saline and methylene blu;
* 1/3 patients will be treated with fluid-filled IGB inflated with 600 ml of saline and methylene blu;
* 1/3 patients will be treated with fluid-filled IGB inflated with 700 ml of saline and methylene blu.

All FF-IGB will be placed into the gastric cavity through the mouth by a gastroscope and filled at the specific volume with 90% of saline and 10% methylene blue solution (in order to diagnose an eventual asymptomatic rupture of the intragastric device), as from indications provided in the package leaflet.

All FF-IGB will last in the stomach for 6 months, as from indications provided in the package leaflet.

An esophagogastroduodenoscopy will be performed 6 months later the endoscopic bariatric procedure for FF-IGB removal.

STATISTICS Sample characteristics will be summarized with means and standard deviations (SD) or medians and 25°-75° percentiles (IQR) for quantitative variables, and absolute and relative (percentages) frequencies for qualitative ones. Shapiro-Wilk test will be used to assess normality of data distribution. Relationship between two quantitative variables will be assessed by calculating Pearson or Spearman correlation coefficients. Pearson Chi Square or Fisher exact tests will be used to evaluate differences of qualitative variables. Differences in quantitative variables between groups will be investigated with unpaired t-test or one-way analysis of variance (ANOVA), or non-parametric methods (Mann-Whitney's and Kruskal-Wallis' tests) if assumptions of parametric tests will not be satisfied.

For post hoc multiple testing, we will adjust the alpha level by using the Bonferroni correction. A p-value less than 0.05 will be considered statistically significant. Jamovi version 2.3 software (The jamovi project, Newcastle, Australia) will be used for statistical computation.

INFORMED CONSENT STATEMENT All patients will be required to give informed consent to the study. All clinical data will be obtained after each patient agreed to treatment by written consent.

DATA RETENTION Data will be retained by the Mater Olbia Hospital in the electronic archive provided for each patient during their first admission at Hospital, as it always happens for all patients.

INSURANCE All patients will be covered by the regular insurance provided by the Mater Olbia Hospital for inpatients and outpatients as the same steps are scheduled also for each patient who should undergo an endoscopic bariatric procedure out of this study.

COSTS No additional costs will be required as at Mater Olbia Hospital the same steps are provided also for each patient who should undergo an endoscopic bariatric procedure out of this study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years, obesity grade I-III, or overweight with at least one obesity-related comorbidity

Exclusion Criteria:

* history of bariatric surgery or endoscopy, allergies to methylene blue, childbearing or not willing to participate or comply with follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Weight loss defined by percentage of Total Weight Loss and Excess Weight Loss | From enrollment to the end of treatment at 6 months
  The primary end point was weight loss defined by percentage of TWL (initial weight minus current weight) / (initial weight) x 100) and percentage EWL (initial weight minus follow-up weight) / (initial weight minus ideal weight for BMI 25) x 100%).

SECONDARY OUTCOMES:
Adverse events (epigastric pain, nausea and vomiting) | From enrollment to the end of treatment at 6 months
  Evaluation of adverse events (epigastric pain, nausea and vomiting, or any other issues (i.e., electrolyte imbalance, chest pain) after intragastric balloon placement requiring additional medical/endoscopic therapy or clinical investigation during hospitalization or until removal)
Early balloon removal | From enrollment to the end of treatment at 6 months
  Detection of early intragastric balloon removal
Improvement of disease specific Quality of Life | From enrollment to the end of treatment at 6 months
  Improvement of disease specific Quality of Life measured by EQ-5D test or Baros test

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore F Vadala di Prampero, Principal Investigator — Mater Olbia Hospital
Locations (1):
- Mater Olbia Hospital, Olbia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar N, Bazerbachi F, Rustagi T, McCarty TR, Thompson CC, Galvao Neto MP, Zundel N, Wilson EB, Gostout CJ, Abu Dayyeh BK. The Influence of the Orbera Intragastric Balloon Filling Volumes on Weight Loss, Tolerability, and Adverse Events: a Systematic Review and Meta-Analysis. Obes Surg. 2017 Sep;27(9):2272-2278. doi: 10.1007/s11695-017-2636-3. PMID 28285471